CLINICAL TRIAL: NCT03049657
Title: Randomized Clinical Trial to Compare the Efficacy of Angiolite Stent Versus a Second-generation Drug-eluting Stent Such as Xience in Patients With Indication of Percutaneous Coronary Intervention
Brief Title: Efficacy of Angiolite Stent vs a Second-generation Drug-eluting Stent Xience for Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiva2 S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ANGIOLITE
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease; Drug-eluting Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANGIOLITE (Active Comparator): Compare the efficacy of Angiolite Stent versus a second-generation drug-eluting stent such as Xience stent.
  Interventions: Device: Angiolite
- Xience (Active Comparator): Compare the efficacy of Angiolite Stent versus a second-generation drug-eluting stent such as Xience stent.
  Interventions: Device: Xience

INTERVENTIONS:
Device: Angiolite — Percutaneous coronary intervention
  Arms: ANGIOLITE
Device: Xience — Percutaneous coronary intervention
  Arms: Xience

SUMMARY:
Clinical trial with an "European Community marked" medical device in patients with ischemic heart disease and clinical indication of coronary revascularization with drug-eluting stent.

Clinical follow-up will be done according to this way: first month telephone or face-to-face interview and at 6 ± 1 month an Angiography follow up + OCT (optical coherence tomography)

A randomized clinical trial to compare the efficacy of Angiolite Stent versus a second-generation drug-eluting stent such as Xience stent.(non-inferiority design)

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical or subclinical ischemic heart disease with indication of percutaneous revascularization.
* "De Novo" lesions ≥ 70%
* Reference diameters ≥ 2 mm and ≤ 4 mm Accepted participation in the registration with the signing of informed consent

Exclusion Criteria:

* Cardiogenic shock
* Pregnancy
* Intolerance or allergy to anti platelet or anticoagulant therapy
* Elective surgical procedure scheduled within 6 months after inclusion in the study
* Expectancy of life of less than 1 year.
* Impossibility of doing 1 year clinical follow-up.
* Primary angioplasty in patients with killip class III-IV or mechanical complications.
* Patient with pre-procedure restenosis.
* Patients who will not be treated all lesions with the Angiolite stent.
* Total occlusions
* Truncus disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Efficacy:Measure the late loss (LL) in the follow-up of the Angiolite stent is not different from the late loss of the xience stent (non-inferiority) | 6 months
  Measure the late loss (LL) in the follow-up of the Angiolite stent is not different from the late loss of the xience stent (non-inferiority)
Safety:Compare TLF rate (cardiovascular death, target vessel-related myocardial infarction (MI) with definite thrombosis or ischemia-driven Target Lesion Revascularization (TLR)) | 1 year
  Compare TLF rate (cardiovascular death, target vessel-related myocardial infarction (MI) with definite thrombosis or ischemia-driven Target Lesion Revascularization (TLR)) during follow-up for no differences between Angiolite and Xience stents

SECONDARY OUTCOMES:
Follow up | 1 year
  Compare differences between Angiolite and Xience stent during the follow-up in independent components of the major adverse cardiac events rate: All cause death, any myocardial infarction and any revascularization
Thrombosis rate | 1 year
  Discard differences in definite and probable thrombosis rate (according to Academic Research Consortium criteria) between both stents Angiolite and Xience
MACE (Major Adverse Cardiac Events) | 1 year
  - Compare the differences between the rate of MACE (all-cause death, any myocardial infarction and any revascularization) of Angiolite and Xience during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ibares, Study Director — Cardiva2 S.L.
Locations (11):
- Spain (11):
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital de León, León, León
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Infanta Cristina, Badajoz
  - Hospital Valle de Hebrón, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital La Paz, Madrid
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No